CLINICAL TRIAL: NCT04851990
Title: A Parallel Pilot Study to Assess the Safety and Tolerability of Long-term Use of Patented Transdermal Patches in Healthy Adults.
Brief Title: Assessment of the Safety & Tolerability of Long-term Use of Patented Transdermal Patches in Healthy Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horopito Limited (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFCRO-135
Record Dates: First submitted 2021-04-13; First posted 2021-04-21 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Vitamin D

STUDY DESIGN:
Intervention Model Description: 2 Arms with 15 Subjects per group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Large Patch (Experimental): To Better Days Large Patch
  1 patch applied daily by 9am - in situ for 24 hours Dosage: vitamin D 30,000 IU + dextrose 13mg
  Interventions: Other: To Better Days Large Patch
- Small patch (Experimental): To Better Days Small Patch
  1 patch applied daily by 9am - in situ for 24 hours Dosage: vitamin D 30,000 IU + dextrose 13mg
  Interventions: Other: To Better Days Small Patch

INTERVENTIONS:
Other: To Better Days Large Patch — Large patch containing vitamin D & Dextrose for transdermal absorption
  Arms: Large Patch
Other: To Better Days Small Patch — Small patch containing vitamin D & Dextrose for transdermal absorption
  Arms: Small patch

SUMMARY:
This is a pilot study to assess the safety and tolerability of long-term use of patented transdermal vitamin D patches in healthy adults.

DETAILED DESCRIPTION:
A randomised, parallel, pilot study to assess the safety and tolerability of long-term use of patented transdermal patches in healthy adults. The study consists of 4 on-site visits: the Screening Visit (Visit 1, Week -2), the Baseline Visit (Visit 2, Week 0), Visit 3 (Week 4), and the End of Intervention Visit (Week 8).

ELIGIBILITY:
Inclusion Criteria:

* 1. Individuals who are willing to participate in the study and comply with its procedures.

  2. Individuals who are able to give written informed consent. 3. Individuals between 18-70 years old. 4. Has a BMI between 18-32 kg/m2 (inclusive). 5. Individuals who are willing to not undertake overseas travel for the duration of the study or engage in excessive sun-exposure or use of sun lamps or tanning beds for the duration of the study.

  6. Individuals who are willing to maintain their current diet and not change supplement usage for the duration of the study.

  7. Individuals who are willing to self-administer finger prick sampling. 8. Individuals who are willing to avoid strenuous exercise or exposing the patch to external sources of direct heat e.g., heating pads or electric blankets, heat lamps, saunas, hot tubs, heated water beds, and prolonged direct sunlight, while wearing the patch.

  9. Individuals willing to refrain from swimming or other sports involving immersion in water for the duration of the study.

  10. Individuals who have Serum 25-Hydroxyvitamin D concentration of ≥15 nmol/L and ≤100 nmol/L at screening.

Exclusion Criteria:

* 1. Are less than 18 or greater than 70 years old. 2. Participants who are pregnant, breastfeeding, or wish to become pregnant during the study.

  3. Individuals currently of childbearing potential, but not using an effective method of contraception, as outlined below:
  1. Complete abstinence from intercourse two weeks prior to administration of Investigational Product, throughout the clinical trial, until the completion of follow-up procedures or for two weeks following discontinuation of the Investigational Product in cases where participant discontinues the study prematurely. (Participants utilising this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit).
  2. Has a male sexual partner who is surgically sterilised prior to the Screening Visit and is the only male sexual partner for that participant.
  3. Sexual partner(s) is/are exclusively female.
  4. Use of acceptable method of contraception, such as a spermicide, mechanical barrier (e.g., male condom, female diaphragm) or contraceptive pill. The participant must be using this method for at least 2 weeks prior to use of the Investigational Product and at least 1 week following the end of the study.
  5. Use of any non-hormonal intrauterine device (IUD) or contraceptive implant with published data showing that the highest expected failure rate is less than 1 % per year. The participant must have the device inserted at least 2 weeks prior to the first Screening Visit, throughout the study, and 2 weeks following the end of the study.

     4. Individuals who are hypersensitive to any of the components of the investigational product.

     5. Individuals who have a condition affecting the integrity of the skin (e.g., psoriasis or eczema).

     6. Individuals who are taking, or have taken, any prescribed or over the counter (OTC) drug and antacids, supplements, or herbal remedies in the 14 days before patch administration including any drugs known to interfere with vitamin D metabolism (e.g., steroids, orlistat, cholestyramine, phenytoin, statins, thiazide diuretics etc.). Occasional use of paracetamol up to a maximum of 2 g per day, hormone replacement therapy [HRT] or hormonal contraception are permissible.

     7. Individuals who have taken calcium supplements within the previous 8 weeks. 8. Individuals who are taking vitamin D supplements greater than 10 micrograms per day.

     9. Individuals with any history of or concurrent clinically significant diseases or conditions (e.g., kidney or liver dysfunction).

     10. Individuals with a known history of allergy to plasters or patches. 11. Individuals who have planned major changes in lifestyle (i.e., diet, dieting, exercise level, travelling) during the duration of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing at least one treatment-emergent adverse event (TEAE) including causality, severity, and seriousness assessments. | Baseline to week 8
  Record number of individual participants experiencing TEAE
Number of treatment-emergent adverse event (TEAE) including causality, severity, and seriousness assessments. | Baseline to 8 weeks
  Record number of TEAE per treatment arm
Number of participants with discontinuations due to AEs or TEAEs | Baseline to 8 weeks
  Record any participants discontinued due to TEAE
Change in Full Blood Count | Baseline to week 8
  Monitor blood safety parameters
Change in blood lipids - total cholesterol, HDL and LDL, triglycerides mmol/l | Baseline to week 8
  Monitor blood safety parameters
Change in Liver Function Tests - IU/l - alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, gama-glutamyl transferase | Baseline to week 8
  Monitor blood safety parameters
Change in blood glucose mmol/l | Baseline to week 8
  Monitor blood safety parameters
Change in blood bilirubin mg/dl | Baseline to week 8
  Monitor blood safety parameters
Change in blood calcium mg/dl | Baseline to week 8
  Monitor blood safety parameters
Change in blood protein g/l - total protein, albumin & globulin | Baseline to week 8
  Monitor blood safety parameters
Change in blood creatine mg/dl | Baseline to week 8
  Monitor blood safety parameters
Change in blood urea mg/dl | Baseline to week 8
  Monitor blood safety parameters
Change in blood uric acid mg/dl | Baseline to week 8
  Monitor blood safety parameters
Change in blood electrolytes mmol/l - sodium, potassium, chloride, bicarbonate, magnesium & phosphate | Baseline to week 8
  Monitor blood safety parameters
Baseline Serum Vitamin D (25-OH) nmol/l | Baseline
  Monitor blood safety parameters
Change in blood pressure - systolic blood pressure (mmHg) & diastolic blood pressure (mmHg) | Baseline to 8 weeks
  Monitor safety measurements
Change in heart rate (BPM) | Baseline to 8 weeks
  Monitor safety measurements
Change in body temperature (˚C) | Baseline to 8 weeks
  Monitor safety measurements

SECONDARY OUTCOMES:
Change in serum vitamin D levels, measured using at-home self-administered finger prick -nmol/l | Baseline - 8 weeks
  Measure change to plasma vitamin D in response to daily patch application

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dinan, Principal Investigator — Atlantia Food Clinical Trials
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jefferson A, Borges C. Evaluation of the safety, tolerability and plasma vitamin D response to long-term use of patented transdermal vitamin D patches in healthy adults: a randomised parallel pilot study. BMJ Nutr Prev Health. 2022 Jul 27;5(2):217-226. doi: 10.1136/bmjnph-2022-000471. eCollection 2022 Dec. PMID 36619342